CLINICAL TRIAL: NCT00109889
Title: A Prospective Observational Study of Patients With Solitary Plasmacytoma Using a Modified Staging System Supplemented by an MRI and Whole Body FDG-PET Scan
Brief Title: S0340 MRI and Fludeoxyglucose F18 PET in Diagnosing Solitary Plasmacytoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CDR0000426422; U10CA032102 (NIH); S0340 (Other: SWOG)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Multiple Myeloma; Plasmacytoma
Keywords: extramedullary plasmacytoma; isolated plasmacytoma of bone
MeSH Terms: conditions — Multiple Myeloma; Plasmacytoma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI and PET (Other): Magnetic resonance imaging and positron emission tomography
  Interventions: Procedure: magnetic resonance imaging; Procedure: positron emission tomography

INTERVENTIONS:
Procedure: magnetic resonance imaging — magnetic resonance imaging (MRI)
  Other Names: MRI
Procedure: positron emission tomography — positron emission tomography (PET)
  Other Names: PET

SUMMARY:
RATIONALE: Diagnostic procedures, such as magnetic resonance imaging (MRI) and fludeoxyglucose F 18 positron emission tomography (^18FDG-PET) may help diagnose solitary plasmacytoma.

PURPOSE: This clinical trial is studying MRI and ^18FDG-PET to see how well they work in diagnosing patients with solitary plasmacytoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the proportion of patients who are misclassified as true solitary plasmacytoma by MRI and whole-body fludeoxyglucose F 18 positron emission tomography as a supplement to imaging with skeletal survey.
* Determine the feasibility of accruing patients to this study.
* Determine, preliminarily, biological correlates and prognostic groups that may relate to progression to symptomatic disease in patients undergoing these imaging procedures.
* Correlate germline genetic polymorphisms with overall clinical course in patients undergoing these imaging procedures.

OUTLINE: This is a multicenter study.

Within 28 days after study entry, patients undergo gadolinium MRI of the head, spine, and pelvis (and other sites, if indicated). Patients then receive fludeoxyglucose F 18 IV followed 90 minutes later by whole-body positron emission tomography (^18FDG-PET) OR whole-body CT scan/PET. Patients with a confirmed diagnosis of solitary plasmacytoma undergo MRI and ^18FDG-PET as above at 1 year and then annually for 10 years in the absence of disease progression (i.e., change of status to solitary plasmacytoma with active myeloma or biopsy confirmed stage IB or higher multiple myeloma).

After completion of study procedures, patients are followed every 6 months for 10 years.

PROJECTED ACCRUAL: A total of 110 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solitary plasmacytoma of 1 of the following types:

  * Solitary bone plasmacytoma
  * Extraosseus solitary plasmacytoma
* Bone marrow plasmacytosis < 10% within the past 4 weeks
* Low serum and/or urine M-protein meeting ≥ 1 of the following criteria:

  * Serum IgG < 3.5 g/dL
  * Serum IgA < 2.0 g/dL
  * Urine M-protein (kappa or lambda) < 1.0 g/24 hours
* No lytic lesions on skeletal survey other than a single lesion associated with solitary plasmacytoma within the past 4 weeks

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin ≥ 10 g/dL* AND/OR
* No hemoglobin 2 g/dL < lower limit of normal* (LLN) NOTE: *Patients with a history of hemoglobin < 10 g/dL AND/OR < 2 g/dL < LLN that has corrected or improved after epoetin alfa but requires continued treatment with epoetin alfa are not eligible

Hepatic

* Not specified

Renal

* Calcium ≤ 10.5 mg/dL OR
* Calcium normal
* Creatinine ≤ 2 mg/dL

Other

* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix or breast, or stage I or II cancer that is currently in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* No prior high-dose steroids except to relieve neurological compromise

Radiotherapy

* Prior localized radiotherapy for myeloma allowed
* Concurrent radiotherapy allowed

Surgery

* Prior surgery for myeloma allowed

Other

* No other prior therapy for myeloma
* Concurrent enrollment in protocol SWOG-S0309 (Myeloma Specimen Repository) allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
proportion of patients misclassified as solitary plasmacytoma | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej J. Jakubowiak, MD, PhD, Study Chair — University of Michigan Rogel Cancer Center; Janet S. Biermann, MD, Study Chair — University of Michigan Rogel Cancer Center; Paul Okunieff, MD, Study Chair — James P. Wilmot Cancer Center
Locations (26):
- United States (26):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Sletten Regional Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming